CLINICAL TRIAL: NCT00806858
Title: NovoPen®4 Clinical Experience Programme: A Multicentre, Observational Study of NovoPen®4 on Treatment Satisfaction of Insulin Therapy in Type 1 or Type 2 Subjects With Diabetes Mellitus
Brief Title: Observational Study of NovoPen® 4 on Treatment Satisfaction of Insulin Therapy in Type 1 or Type 2 Subjects With Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: MS236-3663
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Device: NovoPen® 4

INTERVENTIONS:
Device: NovoPen® 4 — Insulin administration by means of a NovoPen® 4 pen device

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate subjects' treatment satisfaction and to evaluate subjects' preference of pen device and the incidence of clinical technical complains while using NovoPen® 4 under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with Type 1 or Type 2 diabetes and accepting to use NovoPen® 4. The selection will be at the discretion of the individual physician.
* A study specific signed informed consent must be signed by each subject before any study-related activities or information is collected, if required by local regulations

Exclusion Criteria:

* Subjects who are unlikely to comply with the protocol, e.g., unwillingness to cooperate, inability to return for the final visit
* Subjects with known or suspected allergy to any insulin or any of its excipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with Type 1 or Type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 526 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The change in subjects' satisfaction with insulin therapy, measured by change from visit 1 to visit 2 in subject treatment satisfaction scores on the DTSQ (Diabetes Treatment Satisfaction Questionnaire) | 3 months

SECONDARY OUTCOMES:
Subjects' device preference | 3 months
Subjects' NovoPen® 4 evaluation | 3 months
Number of clinical technical complaints | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com